CLINICAL TRIAL: NCT02032251
Title: Reduction of Sperm DNA Fragmentation by Oral Ginger (Zingiberofficinale) Extract Treatment
Brief Title: Reduction of Sperm DNA Fragmentation by Oral Ginger
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: royan-Emb-017
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2009-10

CONDITIONS: Infertility
Keywords: Sperm DNA damage ejaculated spermatozoa Ginger Herbal Drug Herbal medicine
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ginger (Experimental): The patients with infertility that underwent oral administration of ginger.
  Interventions: Drug: oral administration of ginger
- Placebo (Placebo Comparator): The patients with infertility that receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral administration of ginger — Oral administration of ginger in patients with infertility.
  Other Names: Administration of herbal drug
  Arms: ginger
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double blind, controlled clinical trials assess the efficacy of the ginger oral treatment on sperm DNA fragmentation, sperm parameters and male hormones.

DETAILED DESCRIPTION:
Sperm DNA fragmentation is known to affect male fertility. Previous findings have suggested the implication of oxidative stress in the etiology of this pathological condition. The present study was designed to find out DNA fragmentation in ejaculated spermatozoa can be reduced by oral treatment with Ginger extract. 71 men with unexplained or Idiopathic infertility were randomized between a Ginger treatment (500 milligram daily for 3months) group and a placebo group.

Sperm DNA fragmentation was evaluated by Terminal deoxyribonucleotidyltransferase-mediated dUTP nick-end labeling assay (TUNEL) before and after treatment. No differences in basic sperm parameters were found between the Ginger treatment and the placebo group before or after treatment. However, the percentage of DNA-fragmented spermatozoa was markedly reduced (P< .005) in the Ginger treatment group after the treatment as compared with the pretreatment values). No difference in the pretreatment and post treatment incidence of sperm DNA fragmentation was observed in the placebo group. These data show that sperm DNA damage can be efficiently treated with oral Ginger extract administered during a relatively short time period.

ELIGIBILITY:
Inclusion Criteria:

* men with idiopathic infertility or unexplained

Exclusion Criteria:

* history of varicocele, genitourinary inflammation or infection
* history of cigarette smoking.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
sperm DNA fragmentation | 3 months
  Evaluation the percent of the reduction of sperm DNA fragmentation 3 months after ginger administration.

SECONDARY OUTCOMES:
male hormones | 3months
  Evaluation the effect of ginger on male hormones 3 months after oral administration.
sperm count | 3 months
  Evaluation the ginger on sperm count 3 months after oral administration.
sperm motility | 3 months
  Evaluation the effect of ginger on sperm motility 3 months after oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Ali DaliriHampa, MD, Study Director — Department of Andrology, Reproductive Biomedicine Center, Royan Institute for Reproductive Biomedicine; Eyed Jalil Hosseini, MD, Study Director — Department of Andrology, Reproductive Biomedicine Center, Royan Institute for Reproductive Biomedicine; Hani Department of Andrology, Reproductive Biomedicine Center, Roya, MSc, Principal Investigator — Department of Andrology, Reproductive Biomedicine Center, Royan Institute for Reproductive Biomedicine
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org